CLINICAL TRIAL: NCT02821546
Title: Aggressive Fluid Hydration for the Prevention of Post-ERCP Pancreatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nonthalee Pausawasdi, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Si416/2014
Record Dates: First submitted 2016-05-27; First posted 2016-07-01 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard hydration (Placebo Comparator): Patients underwent first-time ERCP to receive standard fluid hydration with Lactated Ringer's solution at a rate calculated by the Holliday-Segar method given peri-procedurally starting 2 hours prior to procedure, and continued during and after procedure to complete 24 hours.
  Interventions: Drug: Lactated Ringer's solution
- aggressive hydration (Active Comparator): Patients underwent first-time ERCP to receive aggressive fluid hydration with Lactated Ringer's solution at a rate of 150 ml/hr starting 2 hours prior to procedure, and continued during and after procedure to complete 24 hours.
  Interventions: Drug: Lactated Ringer's solution

INTERVENTIONS:
Drug: Lactated Ringer's solution — Standard fluid hydration with Lactated Ringer's solution is calculated based on Holiday Segar's equation Aggressive hydration with Lactated Ringer's solution is defined as administration of 150 ml/hour of fluid
  Other Names: Ringer's Lactated solution

SUMMARY:
Aggressive hydration with lactated Ringer's solution (LRS) has been shown in a preliminary research to reduce the incidence of post-endoscopic retrograde cholangiopancreatography (ERCP) pancreatitis. This randomized, controlled trial was designed to assess the effect of peri-procedural aggressive intravenous hydration with LRS on the incidence of post ERCP pancreatitis.

DETAILED DESCRIPTION:
Patients underwent first-time ERCP were randomly assigned (1:1) to receive either LRS at a rate of 150 ml/hr starting 2 hours prior to procedure, and continued during and after procedure to complete 24 hours (aggressive hydration) or LRS at a rate calculated by the Holliday-Segar method given peri-procedurally as described earlier (standard hydration). Visual analog scale, serum amylase, lipase, C-reactive protein (CRP), and urine analysis were assessed prior to procedure and 24 hours after. The primary endpoint was post ERCP pancreatitis defined as new or increased epigastric pain persisting for ≥24 hours, elevation of amylase or lipase >3 times the upper limit of normal.

ELIGIBILITY:
Inclusion Criteria:

* patients at age between 18-65 years old undergoing first time ERCP

Exclusion Criteria:

* Ongoing acute pancreatitis
* Chronic pancreaittis
* Prior sphincterotomy
* Ongoing hypotension including those with sepsis
* Cardiac insufficiency (CI, >NYHA Class II heart failure)
* Renal insufficiency (RI, creatinine clearance <40mL/min)
* Severe liver dysfunction (albumin < 3mg/dL)
* Respiratory insufficiency (defined as oxygen saturation < 90%)
* Pregnancy
* Hyponatremia (Na+ levels < 130mEq/L))
* Hypernatremia (Na+ levels > 150mEq/L)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2014-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
post ERCP pancreatitis | 24 hours
  Post ERCP pancreatitis is defined as hyperamylasemia (amylase >3 times the upper limit of normal [300 U/L]) and pancreatic pain (epigastric abdominal pain radiating to the back scored by patient as development of or increase of pain ≥3 on a 0-10 visual analogue pain scale and persisting for ≥24 hours after ERCP). In those who had pain before the procedure, pancreatic pain is defined as an increase of ≥3 on the 0-10 visual analogue scale.

SECONDARY OUTCOMES:
severity of post ERCP pancreatitis | 24 hours
  severity is defined by length of hospital stay, mild pancreatitis is defined by hospitalization of 48 hours, moderate pancreatitis is defined by hospitalization of more than 48 hours without additional intervention, severe pancreatitis is defined by hospitalization of greater than 72 hours and/or requiring intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nonthalee Pausawasdi, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elmunzer BJ, Scheiman JM, Lehman GA, Chak A, Mosler P, Higgins PD, Hayward RA, Romagnuolo J, Elta GH, Sherman S, Waljee AK, Repaka A, Atkinson MR, Cote GA, Kwon RS, McHenry L, Piraka CR, Wamsteker EJ, Watkins JL, Korsnes SJ, Schmidt SE, Turner SM, Nicholson S, Fogel EL; U.S. Cooperative for Outcomes Research in Endoscopy (USCORE). A randomized trial of rectal indomethacin to prevent post-ERCP pancreatitis. N Engl J Med. 2012 Apr 12;366(15):1414-22. doi: 10.1056/NEJMoa1111103. PMID 22494121
- [Background] Buxbaum J, Yan A, Yeh K, Lane C, Nguyen N, Laine L. Aggressive hydration with lactated Ringer's solution reduces pancreatitis after endoscopic retrograde cholangiopancreatography. Clin Gastroenterol Hepatol. 2014 Feb;12(2):303-7.e1. doi: 10.1016/j.cgh.2013.07.026. Epub 2013 Aug 3. PMID 23920031
- [Background] Adler DG, Baron TH, Davila RE, Egan J, Hirota WK, Leighton JA, Qureshi W, Rajan E, Zuckerman MJ, Fanelli R, Wheeler-Harbaugh J, Faigel DO; Standards of Practice Committee of American Society for Gastrointestinal Endoscopy. ASGE guideline: the role of ERCP in diseases of the biliary tract and the pancreas. Gastrointest Endosc. 2005 Jul;62(1):1-8. doi: 10.1016/j.gie.2005.04.015. No abstract available. PMID 15990812
- [Derived] Chang A, Pausawasdi N, Charatcharoenwitthaya P, Kaosombatwattana U, Sriprayoon T, Limsrivilai J, Prachayakul V, Leelakusolvong S. Continuous Infusion of Fluid Hydration Over 24 Hours Does Not Prevent Post-Endoscopic Retrograde Cholangiopancreatography Pancreatitis. Dig Dis Sci. 2022 Aug;67(8):4122-4130. doi: 10.1007/s10620-021-07256-z. Epub 2021 Oct 15. PMID 34655014